CLINICAL TRIAL: NCT04189978
Title: Study of the Impact of Microbial Exposure of the Habitat at the Time of Birth on the Development of Allergic Diseases.
Brief Title: Impact of Microbial Exposure of the Habitat at the Time of Birth on the Development of Allergic Diseases.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Michel, Head of immuno-allergology departement, Brugmann University Hospital
Other Study IDs: CHUB-ENVIBRU
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Allergic Disorder
MeSH Terms: conditions — Hypersensitivity | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2001-2002 study participants: Children who participated in the study conducted in 2001-2002, their parents and the siblings who were exposed to the same environment at this period.
  Interventions: Diagnostic Test: Clinical evaluation

INTERVENTIONS:
Diagnostic Test: Clinical evaluation — The assessment is based on a comprehensive questionnaire, a simple clinical examination, an spirometry test, allergic skin tests, measurement of the exhaled fraction of NO (FeNO) and blood serum analysis.

SUMMARY:
In 2001-2002, a longitudinal study on the risk of atopic sensitization in children was conducted by the Pneumo-Allergology and Pediatrics departments of the CHU Saint-Pierre Hospital and at the Neonatology Department of the Queen Fabiola Children's University Hospital (HUDERF). The aim of the study was to study bacteria and endotoxins in airborne dust in Brussels homes in order to evaluate their impact on the development of allergic diseases in newborns.

Between December 2000 and August 2002, 114 children (67 from HUDERF and 47 from CHU St-Pierre) were included in the study. These were eutrophic children without acquired pathology or known genetics.

Simultaneously a microbial habitat assessment was performed based on a detailed description and on endotoxin assays in the airborne and deposited dust (mainly mattress).These data can be used to define habitats with high or low contamination.Samples for microbial analyzes (Gram positive and negative and mold) were also carried out.

Preliminary results suggested:

1. A protective effect of airborne dust endotoxins on the risk of developing atopic dermatitis in children at 6 and 12 months of life,
2. An effect of endotoxins promoting the occurrence of wheezing in children after 6 months.

In this current, new study, the investigators will recontact the children who were included in the 2003 study. The goal is to evaluate them clinically and allergically and associate the risk of sensitization / allergic diseases with the microbial exposure of the habitat, measured during the neonatal period.

Siblings and parents who were exposed during the same period will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Children who participated in the study conducted in 2001-2002, their parents and the siblings who were exposed to the same environment at this period.

Exclusion Criteria:

None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children who participated in the study conducted in 2001-2002, their parents and the siblings who were exposed to the same environment at this period.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of positivity of allergic skin tests | 1 year
  Prevalence of positivity of allergic skin tests
Prevalence of positivity of ImmunoCAP tests | 1 year
  Prevalence of positivity of ImmunoCAP tests

SECONDARY OUTCOMES:
Prevalence of clinical manifestations of allergy | 1 year
  Prevalence of clinical manifestations of allergy (atopic eczema, food allergy, asthma and rhinitis).
Prevalence of confirmed asthma | 1 year
  Prevalence of confirmed asthma (clinical manifestations, spirometry and FeNO)
Spirometry results | 1 year
  Spirometry results
Exhaled fraction of NO (FeNO) results | 1 year
  Exhaled fraction of NO (FeNO) results
Eosinophilia count | 1 year
  Eosinophilia count
Socio-cultural status | 1 year
  Socio-cultural status

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Michel, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No